CLINICAL TRIAL: NCT00242697
Title: A Randomized Double-Blind Comparison of Combined General-Spinal Anesthesia to General Anesthesia for Coronary Artery Surgery
Brief Title: Double-Blind Comparison of Combined General-Spinal Anesthesia to General Anesthesia for Coronary Artery Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARF1
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2005-10

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Surgery
Keywords: coronary artery bypass surgery; anesthesia, general; anesthesia, spinal; heart-lung machine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Anesthesia

INTERVENTIONS:
Procedure: spinal analgesia and anesthesia for coronary artery surgery

SUMMARY:
Use of neuraxial agents in anesthesia for cardiac surgery is expanding. We have used combined general-spinal anesthesia for cardiac surgery for 12 years. We hypothesized that compared to general anesthesia, the combined techniques would provide comparable intraoperative hemodynamics and improved postoperative analgesia. This study subjected these techniques to a double-blind randomized trial.

DETAILED DESCRIPTION:
Use of neuraxial agents in anesthesia for cardiac surgery is expanding. We have used combined general-spinal anesthesia for cardiac surgery for 12 years. We performed a trial in order to determine if our clinical impressions of the techniques would be confirmed. We hypothesized that compared to general anesthesia, the combined techniques would provide comparable intraoperative hemodynamics and improved postoperative analgesia. This study subjected these techniques to a double-blind randomized trial.

METHODS

After IRB approval, 63 consenting patients undergoing non-emergent coronary artery bypass grafting (CABG) entered a randomized, double-blind trial. Patients received lorazepam 0.03 mg/kg preoperatively, and midazolam 0.03 mg/kg during line insertion and induction. Spinal procedures, performed by an unblinded study anesthesiologist, preceded general anesthesia, which was induced with propofol and rocuronium, and maintained with isoflurane through CPB, and propofol thereafter. All caregivers were blinded to group assignment. Opioid and spinal management defined 3 groups:

GA: Sufentanil IV: 3 μg/kg induction, 1 μg/kg x 2 prn; mock spinal SO: Sufentanil IV: 0.2 μg/kg induction, 0.1 μg/kg x 2 prn; Spinal: sufentanil 50 μg, morphine 0.5 mg, hyperbaric SL: Sufentanil IV: 0.2 μg/kg induction, 0.1 μg/kg x 2 prn; Spinal: sufentanil 25 μg, morphine 0.5 mg, bupivacaine 9.75 mg, hyperbaric

When patients were stable in ICU, propofol was stopped and an extubation protocol begun. Patients received scheduled NSAID and prn opioid, IV or PO. The chi-square test and ANOVA using the Scheffe method for multiple comparisons were applied appropriately.

The primary end points of the study were analgesic requirements, visual analogue pain scores, and duration of endotracheal intubation in the intensive care unit. Secondary endpoints were intraoperative hemodynamic variables, blood catecholamine and lactate levels, anesthetic supplementation, and vasoactive drug support.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing non-emergent primary coronary artery bypass grafting using cardiopulmonary bypass

Exclusion Criteria:

* < 25 or > 80 years of age
* left ventricular ejection fraction < 35%
* receiving inotropic or intraaortic balloon therapy at time of surgery
* receiving intravenous heparin therapy at time of surgery
* pre-existing back problems in the lumbar area
* clinical or laboratory evidence of coagulopathy

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 2002-04; Study Completion 2003-07

PRIMARY OUTCOMES:
analgesic requirement in the intensive care unit
visual analogue pain scores in the intensive care unit
duration of endotracheal intubation in the intensive care unit

SECONDARY OUTCOMES:
intraoperative hemodynamic variables
intraoperative blood catecholamine and lactate levels
intraoperative anesthetic supplementation
intraoperative vasoactive drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Charles L MacAdams, MD FRCPC, Principal Investigator — Department of Anesthesia, Foothills Medical Centre, University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] MacAdams, CL et al. Combined general-spinal vs spinal anesthesia for coronary artery bypass grafting. Can J Anesth 73(Suppl I):A73,2003.